CLINICAL TRIAL: NCT04103801
Title: Substance P as a Biomarker to Evaluate the Reduction of Multiple Immunization Pain Among Infants and Toddlers: A Randomized Controlled Trial
Brief Title: Substance P as a Biomarker to Evaluate the Reduction of Multiple Immunization Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 127-2015
Record Dates: First submitted 2018-10-17; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Immunisation Anxiety Related Reaction; Pain, Acute
Keywords: Sucrose,; Substance P,; Pain,; Immunization.
MeSH Terms: conditions — Acute Pain; Pain | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrose group (Experimental): This group received the 2 ml of sweet solution (sucrose)
  Interventions: Dietary Supplement: Sucrose
- Water group (Placebo Comparator): This group received the 2 ml of water
  Interventions: Dietary Supplement: Sucrose

INTERVENTIONS:
Dietary Supplement: Sucrose — Participants in the intervention group were given 2 ml dose of 50% sucrose solution and participants in the placebo group were given 2 ml dose of sterile water. Both groups were administered slowly over 30 seconds sublingually via needle-less syringe immediately prior to the immunization injections.
  Other Names: Sweet solution

SUMMARY:
Immunization is one of the most significant preventive health measures in reducing morbidity and mortality caused by infectious diseases. Studies have shown that Sucrose is recommended to reduce pain associated with vaccination in neonates. The main aim of the study was to determine the effectiveness of sucrose in reducing infant's pain outcomes during immunization among 10-24 month-old infants and toddlers.

ELIGIBILITY:
Inclusion Criteria:

* All healthy children who were attending immunization clinic to have their 10-24 month immunization were invited to this study

Exclusion Criteria:

* Exclusion criteria included children: whose parents choose to breastfeed during immunization, who have received an analgesia in the previous 24 hours including Paracetamol (so as not to affect the response to painful stimuli during immunization), who cannot receive their immunization due to the presence of immunization risk factors as determined by the immunization nurse, who are not able to receive a sugar solution, and whose parents refuse to participate.

Ages: 10 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
MBPS | Change MBPS score from the start of injection and up to 3 minutes after immunization
  Modified Behavioral Pain Scale (MBPS) is a validated procedural uni-dimensional pain measurement tool that used to measure behavioral pain outcomes.

SECONDARY OUTCOMES:
Substance P (SP) | Change SP level from the start of injection and up to 3 minutes after immunization
  Change SP level as an indicator of pain and distress level. Saliva was collected from both intervention and placebo groups immediately after treatment in the same manner and similar time schedule. Saliva specimens was immediately cooled in ice and centrifuged at 10,000g at 4 C for 15 min to obtain the supernatant.

OTHER OUTCOMES:
Total crying time | From start of injection and up to 3 minutes after the immunization
  The total crying time duration in minute was measured (using the video) from start of injection and to post-immunization Crying

CONTACTS AND LOCATIONS:
Overall Officials: Manal K, PhD, Principal Investigator — Jordan Uinversity of Sceince and Technology
Locations (1):
- Maternal and child health centers, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
The data is confidential and could not be shared.